CLINICAL TRIAL: NCT06418659
Title: A Clinical Trial Assessing the Safety and Efficacy of Intravenous CD-801 for the Treatment of Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Clinical Trial Evaluating the Safety and Efficacy of Intravenous CD-801 in Treating Advanced HCC Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Wei-Fen Xie, Director, Department of Gastroenterology, Changzheng Hospital, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZXH-HCC-2024-IIT
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Hepatocyte nuclear factor 4α
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: The subjects with advanced HCC will be treated by CD-801 intravenously via a peripheral vein.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD-801 treatment (Experimental): The subjects with advanced HCC will be treated by CD-801 intravenously via a peripheral vein.
  According to Amendment 1, the HNF4α srRNA preparation CD-801 used in the original protocol will expire on December 31, 2024. For participants receiving treatment after this date, the preparation will be switched to CD-GA-102, with the treatment dose converted on a 1:1 basis.
  Interventions: Drug: CD-801

INTERVENTIONS:
Drug: CD-801 — CD-801 will be administered intravenously for the treatment of HCC. The dosing regimen is planned for a second dose 14 ± 3 days post-initial treatment, followed by subsequent treatments every 28 ± 7 days, with adjustments made based on patient tolerance and therapeutic response.
  According to Amendment 1, patients who have received at least 4 cycles of HNF4α srRNA (CD-801 or CD-GA-102) therapy and have a tumor assessment of SD (stable disease) or PD (progressive disease) per mRECIST criteria may, after a comprehensive evaluation by the investigator considering the patient's treatment history and the current safety and efficacy data of HNF4α srRNA, continue HNF4α srRNA at the same dose, or have their dose adjusted, in combination with immunotherapy, targeted therapy, or chemotherapy.

SUMMARY:
The goal of this investigator-initiated, a single-arm, open-label, pilot study is to investigate the safety, tolerability, and efficacy of Intravenous CD-801 treatment in subjects with advanced hepatocellular carcinoma(HCC).

Condition of disease: advanced hepatocellular carcinoma.

Intervention： CD-801 will be administered intravenously for the treatment of HCC. The dosing regimen is planned for a second dose 14 ± 3 days post-initial treatment, followed by subsequent treatments every 28 ± 7 days, with adjustments made based on patient tolerance and therapeutic response. The trial is structured in two phases: dose escalation and dose expansion.

Dose Escalation Phase:

The study employs a i3+3 design to assess escalating CD-801 dosages: 25 μg, 50 μg, and 100 μg. Post-initial dose, a 14-day DLT observation will evaluate tolerability and safety, guiding dose adjustments or selection of the Recommended Dose (RD) for the expansion phase. Cohorts may include up to 9 participants, adjusted for safety.

Dose Expansion Phase:

The expansion phase will use the safe dosage and regimen from the escalation phase, with treatments starting 14 ± 3 days after the initial dose, then every 28 ± 7 days, adjusted as needed. It ends upon complete response, disease progression, toxicity, withdrawal, loss to follow-up, new oncological treatments, or investigator termination, with a final assessment 14 days post-last dose. The phase plans to enroll about 10 participants to further assess CD-801's safety, tolerability, and antitumor effects using mRECIST.

Drug: CD-801, a drug specifically designed to target liver cancer cells and facilitate the expression of HNF4α.

According to Amendment 1, in these two phases, patients who have received at least 4 cycles of HNF4α srRNA (CD-801 or CD-GA-102) therapy and have a tumor assessment of SD (stable disease) or PD (progressive disease) per mRECIST criteria may, after a comprehensive evaluation by the investigator considering the patient's treatment history and the current safety and efficacy data of HNF4α srRNA, continue HNF4α srRNA at the same dose, or have their dose adjusted, in combination with immunotherapy, targeted therapy, or chemotherapy.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the most common form of liver cancer. Recent advancements in understanding tumor biology and the tumor microenvironment, along with the approval of systemic therapeutic agents, including immunotherapy and vascular endothelial growth factor (VEGF)-targeted agents, have dramatically transformed the treatment landscape for advanced stage HCC. However, the survival for advanced HCC patients still remains unsatisfactory.

Differentiation therapy in oncology is defined as a therapeutic strategy that reactivates endogenous differentiation programs and reverts malignant phenotypes. Its hallmark success is the treatment of acute promyelocytic leukemia (APL) by the combination of all-trans retinoic acid (ATRA) and arsenic. Unfortunately, this approach has achieved limited success in solid tumors.

Hepatocyte nuclear factor 4α (HNF4α) is a transcription factor (TF) belonging to the nuclear receptor family. HNF4α is highly enriched in mature hepatocytes and serves as a master regulator of hepatocyte differentiation and hepatic metabolism. Previous studies, including our own and others, have demonstrated that the reduced expression of HNF4α plays a critical role in hepatocarcinogenesis. Restoring HNF4α expression induces the differentiation of HCC cells into mature hepatocytes and has shown significant therapeutic effects in various animal models of HCC.

In this study, the investigators developed CD-801, a drug specifically designed to target liver cancer cells and facilitate the expression of HNF4α, for the treatment of HCC patients. Preclinical studies have shown that CD-801 effectively inhibits the growth of subcutaneous and orthotopic liver tumors in mice. Acute toxicity tests in Sprague-Dawley rats have demonstrated that a single intravenous injection of CD-801 injection at a dose of 150 μg/animal is well-tolerated, with no significant toxicity, indicating good safety profiles.

This trial, structured in two phases: dose escalation and dose expansion, is a single-arm, open-label, exploratory clinical study aimed at evaluating the efficacy, safety, and tolerability of CD-801 administered intravenously through a peripheral vein in the treatment of advanced-stage HCC. The treatment schedule is planned for a second dose 14 ± 3 days post-initial treatment, followed by subsequent treatments every 28 ± 7 days, with adjustments made based on patient tolerance and therapeutic response.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged 18 years or older.
2. Subjects must have confirmed diagnosis of HCC with any of the following criteria according to the American Association for the Study of Liver Diseases criteria.
3. Unresectable HCC.
4. Subjects were not eligible for locoregional or systemic therapies, or had disease progression, or would not benefit after at least one of the conventional therapies.
5. According to mRECIST, subjects should be with at least 1 measurable target lesion.
6. Life expectancy of 12 weeks or more.
7. Subjects must have an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 2.
8. Males with fertility and females of childbearing potential are willing to use a highly effective method of contraception for the entire study period and for 6 months after study drug discontinuation. Females of childbearing age, including premenopausal females and within 2 years after menopause, must have a negative serum pregnancy test result within 7 days prior to the first dose of study treatment.
9. Subjects who had a voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.

Exclusion Criteria:

1. Inadequate liver function：Albumin (ALB) < 25 g/L, or total bilirubin > 5 × the upper limit of normal (ULN), or aspartate aminotransferase (AST), alkaline phosphatase (ALP), or alanine aminotransferase (ALT) >10 × ULN.
2. Inadequate renal function defined as creatinine >1.5 × ULN or calculated creatinine clearance < 40 mL/min.
3. Absolute neutrophil count (ANC) < 1.0×109/L, or Platelets < 30×109/L, or Hemoglobin < 8.5 g/dL.
4. International Normalized Ratio (INR) > 2.3.
5. Subjects with a history of liver transplantation.
6. Subjects with poorly controlled hypertension, diabetes or other serious heart or lung diseases, or with serious dysfunction.
7. Subjects with extrahepatic metastasis who had not received first-line systemic therapies (excluding those who are not eligible for systemic therapies) or who were receiving effective systemic therapy currently.
8. Subjects who had prior anticancer treatment with any locoregional therapies, antiangiogenic targeted therapies, immune checkpoint inhibitors or chemotherapy (within 4 weeks, or within 2 weeks in case of sorafenib), radiotherapy (within 3 weeks), or active traditional Chinese medicine (within 2 weeks) before the first dose of study treatment, except for the treatments after which the disease still progressed according to mRECIST.
9. All toxicities related to prior locoregional or systemic anti-tumor treatments are still grade 2 or more (except for hair loss and other events that have been judged tolerable by researchers).
10. Subjects with complication histories of liver cirrhosis or HCC such as gastrointestinal hemorrhage, overt hepatic encephalopathy, or refractory ascites within 2 weeks prior to the first dose of study treatment.
11. Uncontrolled active infection (eg, lung infections, or abdominal infections).
12. History of malignancy other than HCC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year overall survival rate > 90%), such as adequately treated early gastric carcinoma, carcinoma in situ of the cervix, non-melanoma skin carcinoma, or localized prostate cancer.
13. HBV DNA greater than 500 copies/mL, or HCV RNA greater than 15 U/mL.
14. Subject is positive for Human Immunodeficiency Virus (HIV).
15. Any subject who is allergic to MRI contrast agents.
16. Pregnant/lactating women, or women who have the possibility of pregnancy.
17. Participation in other investigational drug trials within 4 weeks prior to initiation of this study treatment.
18. Any medical or other condition which, in the opinion of the investigator, would preclude participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-10-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
(Escalation part) To evaluate the tolerability and safety for intravenous CD-801 in subjects with hepatocellular carcinoma (HCC) | Through study completion, an average of 2 years
  Safety and tolerability are assessed based on the incidence of Dose-Limiting Toxicities (DLTs) within 14 days post-initial drug administration, along with the frequency and severity of adverse events (AEs), serious adverse events (SAEs), and events leading to treatment discontinuation throughout the treatment period, all evaluated using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
  According to Amendment 1, the primary endpoint has been amended from assessing the incidence and severity of DLTs, adverse events (AEs), serious adverse events (SAEs), and AEs leading to treatment discontinuation (evaluated per NCI-CTCAE 5.0) with HNF4α srRNA therapy to assessing these outcomes for both HNF4α srRNA monotherapy and combination therapy.
(Expansion part) To assess the objective response rate (ORR) by modified Response Evaluation Criteria in Solid Tumours (mRECIST). | From the first study dose date until the date of documented complete response or partial response, assessed up to 24 months
  To assess the proportion of subjects who have best overall response of complete response or partial response at the time of data cutoff based on mRECIST.
  According to Amendment 1, the primary endpoint has been updated from evaluating the ORR per mRECIST with HNF4α srRNA therapy to evaluating the ORR for both monotherapy and combination therapy with HNF4α srRNA per mRECIST.

SECONDARY OUTCOMES:
(Escalation part) To assess the objective response rate (ORR) by mRECIST and RECIST v1.1. | From the first study dose date until the date of documented complete response or partial response, assessed up to 24 months.
  To assess the proportion of subjects who have best overall response of complete response or partial response at the time of data cutoff based on mRECIST and RECIST v1.1.
  According to Amendment 1, this outcome has been updated from evaluating the ORR per mRECIST with HNF4α srRNA therapy to evaluating the ORR for both monotherapy and combination therapy with HNF4α srRNA per mRECIST and RECIST v1.1.
(Expansion part) To evaluate the tolerability and safety for intravenous CD-801 in subjects with HCC | Through study completion, an average of 2 years
  To assess the frequency and severity of AEs, SAEs, and events leading to treatment discontinuation throughout the treatment period, all evaluated using CTCAE 5.0.
  According to Amendment 1, this outcome has been amended from assessing the incidence and severity of DLTs, adverse events (AEs), serious adverse events (SAEs), and AEs leading to treatment discontinuation (evaluated per NCI-CTCAE 5.0) with HNF4α srRNA therapy to assessing these outcomes for both HNF4α srRNA monotherapy and combination therapy.
(Expansion part) The objective response rate based on RECIST v1.1 | From the first study dose date until the date of documented complete response or partial response, assessed up to 24 months
  To assess the proportion of subjects who have best overall response of complete response or partial response at the time of data cutoff based on RECIST v1.1 According to Amendment 1, this outcome has been updated from evaluating the ORR per mRECIST with HNF4α srRNA therapy to evaluating the ORR for both monotherapy and combination therapy with HNF4α srRNA per mRECIST.
Duration of response based on mRECIST and RECIST v1.1 | up to 24 months
  To assess the time from the first documentation of complete response or partial response to the date of first documentation of disease progression or death (whichever occurs first) based on mRECIST and RECIST v1.1
Progression-free survival based on mRECIST and RECIST v1.1 | up to 24 months
  To assess the time from the first study dose date to the date of first documentation of disease progression or death(whichever occurs first) based on mRECIST and RECIST v1.1
Time to progression based on mRECIST and RECIST v1.1 | up to 24 months
  To assess the time from the first study dose date to the date of first documentation of disease progression based on mRECIST and RECIST v1.1
Time to response based on mRECIST and RECIST v1.1 | up to 24 months
  To assess the time from the date of first study dose to the date of first documentation of complete response or partial response based on mRECIST and RECIST v1.1
Disease control rate based on mRECIST and RECIST v1.1 | up to 24 months
  To assess the proportion of subjects who have best overall response of complete response or partial response or stable disease (minimum duration from the initial treatment to stable disease ≥5 weeks) based on mRECIST and RECIST v1.1
Clinical benefit rate based on mRECIST and RECIST v1.1 | up to 24 months
  To assess the proportion of subjects who have best overall response of complete response or partial response or durable stable disease (duration of stable disease ≥ 23 weeks) based on mRECIST and RECIST v1.1
Overall Survival | Throughout the entire course of treatment until the end of the follow-up period, an average of 2 years
  To assess the time from the first study dose date until date of death from any cause . Subjects who are lost to follow-up and the subjects who are alive at the date of data cutoff will be censored at the date the subject was last known alive or the cut-off date, whichever comes earlier.

OTHER OUTCOMES:
Health Related Quality of Life based on the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30). | Through study completion, an average of 2 years
  To evaluate the impact of CD-801 treatment on Health Related Quality of Life for subjects treated using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30).
Health Related Quality of Life based on HCC-specific EORTC QLQ-HCC18 questionnaire. | Through study completion, an average of 2 years
  To evaluate the impact of CD-801 treatment on Health Related Quality of Life for subjects treated using HCC-specific EORTC QLQ-HCC18 questionnaire.
Health Related Quality of Life based on European Quality of Life questionnaire. | Through study completion, an average of 2 years
  To evaluate the impact of CD-801 treatment on Health Related Quality of Life for subjects treated using European Quality of Life questionnaire.
The impact of CD-801 treatment on tumor biomarkers in serum. | Through study completion, an average of 2 years
  To investigate the changes in serum tumor biomarkers among subjects with advanced HCC following CD-801 treatment.
The impact of CD-801 treatment on cytokines in serum. | Through study completion, an average of 2 years
  To investigate the changes in serum cytokines among subjects with advanced HCC following CD-801 treatment.
The impact of CD-801 treatment on immune cell profiling in serum. | Through study completion, an average of 2 years
  To investigate the changes of immune cell profiling in serum among subjects with advanced HCC following CD-801 treatment.
The impact of CD-801 treatment on tumor histopathology. | Through study completion, an average of 2 years
  To investigate the changes of histopathology in tumor tissue among subjects with advanced HCC following CD-801 treatment.
The impact of CD-801 treatment on tumor metabolism. | Through study completion, an average of 2 years
  To investigate the changes of tumor metabolism through metabolomic analysis of liver cancer tissue among subjects with advanced HCC following CD-801 treatment.
The impact of CD-801 treatment on gene expression profiles within tumors. | Through study completion, an average of 2 years
  To investigate the changes of tumor gene expression profiles through next-generation sequencing and single-cell sequencing analysis of liver cancer tissue among subjects with advanced HCC following CD-801 treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Fen Xie, M.D., Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Changzheng Hospital, Shanghai, Shanghai Municipality, China